CLINICAL TRIAL: NCT06938698
Title: PROMs From GEstIC Heart Failure Patients - PROFIC-HF Study
Brief Title: PROMs From GEstIC Heart Failure Patients
Acronym: PROFIC-HF
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar do Porto (Other)
Collaborators: Promptly Health (Industry); EIT Health (Other)
Responsible Party: Principal Investigator, Irene Marques, Internal Medicine Senior Consultant, Centro Hospitalar do Porto
Other Study IDs: 2020.032
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Patient-Reported Outcome Measures; Clinical Outcomes; Quality of Life; Telemedicine; Feasibility Studies
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Heart Failure patients: Patients of the GEstIC Heart Failure clinic will use a digital PROMs system, collecting information on the consultation waiting room and/or with the patient at home using a web based application that runs on the smartphone or computer with internet connection.
  Interventions: Other: PROM collection

INTERVENTIONS:
Other: PROM collection — PROM collection using a digital health web application. PROMs will be based on the HF Standard Set created by the International Consortium of Health Outcomes Measurements (ICHOM), adapted to the patient follow-up protocol already in use by GEstIC. Half the participants will complete the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) and the other half will complete the Minnesota Living with Heart Failure Questionnaire (MLHFQ).

SUMMARY:
Heart failure (HF) is a chronic condition with substantial morbidity, and understanding its effects on patients' quality of life is essential.

Patient-reported outcomes (PROs) are any result of a disease or treatment that comes directly from the patient, without any interpretation from clinicians, using standardized scientifically-validated medical questionnaires, PROMs. Patient-reported outcome measures (PROMs) are the tools used to capture PRO information usually in the form of questionnaires.

The PROMs from GEstIC Heart Failure Patients (PROFIC-HF) study aims to assess the feasibility of digitally recording Patient-Reported Outcome Measures (PROMs) at home in real-world patients enrolled in a multidisciplinary heart failure clinic. Two HF-specific PROMs - Kansas City Questionnaire (KCCQ-12) and the Minnesota Living with Heart Failure Questionnaire (MLHFQ) - and a 2 PROMs for anxiety and depression assessment - Patient Health Questionnaire -2 (PHQ-2) and The Hospital Anxiety and Depression Scale (HADS) will be collected remotely using a digital platform that can be accessed online using a smartphone or a computer.

This study will also evaluate the correlation between quality of life changes (measured by Kansas City Cardiomyopathy Questionnaire (KCCQ-12) versus Minnesota Living with Heart Failure Questionnaire) and changes in clinical reported outcomes: assess the quality of life of real world HFpatients followed in a multidisciplinary heart failure clinic and quantify the impact of hospitalization events on patients' quality of life.

DETAILED DESCRIPTION:
PROFIC-HF will randomize 75 participants to complete the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) and 75 to complete the Minnesota Living with Heart Failure Questionnaire (MLHFQ).

The trial will pilot the use of the digital PROMs system, collected from the consultation waiting room and/or with the patient at home.

PROMs will be based on the HF Standard Set created by the International Consortium of Health Outcomes Measurements (ICHOM), adapted to the patient follow-up program already in use by GEstIC.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent (IC) signed before any study- specific procedure,
* Adult patients diagnosed with HF, undergoing treatment at GEstIC,
* Ability and willingness to understand the proposed questionnaires, per physician judgment and
* Ability and willingness to access the platform for completing the data by themselves or with the help of a caregiver (proxy)

Exclusion Criteria:

* Inability to give the answers to the questions in the questionnaires,
* Moderate or severe cognitive impairment that precludes the understanding of the questions, per physician judgment,
* Malignancy or other non-cardiac condition limiting life-expectancy to < 12 months, per physician judgment or
* Any other condition or therapy that would make the subject unsuitable to this study and would not allow participation for the full planned study period, in the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with Heart Failure, undergoing treatment at GEstIC. Eligible patients will be identified by GEstIC physicians/investigators in HF hospital appointments.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life as measured by KCCQ-12 versus MLHFQ | Measurement at 0, 1 and 6 months after informed consent.
  Kansas City Cardiomyopathy Questionnaire (KCCQ-12) and Minnesota living with Heart Failure (MLHFQ) are a quality of life (QoL) questionnaires specific for heart failure. Patients will be randomized to answer to only one of the questionnaires.
  KCCQ consists of 12 questions specific to HF and appraises QoL over the last two weeks; scores range from 0 to 100, where higher score means better QoL. The MLHFQ consists of 21 questions and appraises QoL over the previous month. Questions are answered using a Likert scale ranging from 0-5; score range is 0-105, with higher score representing a poorer QoL.

SECONDARY OUTCOMES:
Correlation between quality of life changes, measured by Kansas City Cardiomyopathy Questionnaire (KCCQ-12) versus Minnesota Living with Heart Failure Questionnaire (MLHFQ), and changes in clinical reported outcomes. | Measurement at 0, 1 and 6 months after informed consent.
  KCCQ-12 and MLHFQ are HF-specific quality of life questionnaires. Patients will either answer to only one of the questionnaires.
Assessment the effect of HF hospitalizations in the quality of life of real world HF patients. | Measurement at 0, 1 and 6 months from discharge.
  Measurement of quality of life after HF hospitalizations, using Kansas City Cardiomyopathy Questionnaire (KCCQ-12) versus Minnesota living with Heart Failure (MLHFQ). Patients will be randomized to answer to only one of the questionnaires.
  KCCQ consists of 12 questions specific to HF and appraises QoL over the two weeks; scores range from 0 to 100, where higher score means better QoL. The MLHFQ consists of 21 questions and appraises QoL over the previous month. Questions are answered using a Likert scale ranging from 0-5; score range is 0-105, with higher score representing a poorer QoL..
Assessment of anxiety and depression by Hospital Anxiety and Depression Scale (HADS) | Measurement at 0, 1 and 6 months after informed consent.
  HADS will be used to assess anxiety and depression. HADS is a 14-item scale, in which all items are rated on a 4-point Likert scale, and scores are 19 computed by summing the scores of each subscale, for anxiety or depression. Scores range from 0 to 20, where higher scores indicate more anxiety or depression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Marques, MD, Principal Investigator — Centro Hospitalar do Porto
Locations (1):
- Centro Hospitalar Universitário do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burns DJP, Arora J, Okunade O, Beltrame JF, Bernardez-Pereira S, Crespo-Leiro MG, Filippatos GS, Hardman S, Hoes AW, Hutchison S, Jessup M, Kinsella T, Knapton M, Lam CSP, Masoudi FA, McIntyre H, Mindham R, Morgan L, Otterspoor L, Parker V, Persson HE, Pinnock C, Reid CM, Riley J, Stevenson LW, McDonagh TA. International Consortium for Health Outcomes Measurement (ICHOM): Standardized Patient-Centered Outcomes Measurement Set for Heart Failure Patients. JACC Heart Fail. 2020 Mar;8(3):212-222. doi: 10.1016/j.jchf.2019.09.007. Epub 2019 Dec 11. PMID 31838032
- [Background] Marques, I., Gomes, C., Viamonte, S., Ferreira, G. e Mendonça, C. 2017. Clínica Multidisciplinar de Insuficiência Cardíaca: Como Implementar. Medicina Interna. 24, 4 (Dez. 2017), 308-317. DOI:https://doi.org/10.24950/rspmi/R58/17/2017.